CLINICAL TRIAL: NCT04894097
Title: Effect of Magnetic Therapy on Pain and Function in Hemplegic Shoulder Pain Patients
Brief Title: Effect of Magnetic Therapy on Pain and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Ibrahim Ahmed Ibrahim Abu Ella, assistant lecturer, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo University
Record Dates: First submitted 2021-05-16; First posted 2021-05-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2023-02

CONDITIONS: Hemiplegia
Keywords: pain thrshold; ROM
MeSH Terms: conditions — Hemiplegia | interventions — Magnetic Field Therapy

STUDY DESIGN:
Intervention Model Description: * The selected patients will be randomly assigned to two equal groups (study group (GI), and control group (GII).
  * The study group (GI) will be treated by magnetic therapy in addition to design physical therapy program.
  * The control group (GII) will be treated by sham magnetic therapy in addition to the same design physical therapy program of (GI).
Who Masked: Participant
Masking Description: The patients in control group will be treated by sham radial extracorporeal shock wave therapy in addition to, the same design physical therapy program. Stimulation will not deliver as the transmitter head will be removed.
  The patients will receive the same frequency of air pressure and
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): Patients will received low frequency high intensity magnetic therapy
  Interventions: Device: magnetic therapy
- control group (Sham Comparator): The patients in this group will be treated by sham magnetic therapy
  Interventions: Device: magnetic therapy

INTERVENTIONS:
Device: magnetic therapy — High intensity low frequency magnetic therapy

SUMMARY:
The purpose of the current study will be focused on the following issues. Evaluation of the effect of magnetic therapy on the pressure pain threshold and disability in stroke hemiplegic shoulder.

DETAILED DESCRIPTION:
Further understanding of rotator cuff tendon impairment and other shoulder soft tissue structural abnormalities in stroke patients may help clinicians in assigning more complete therapeutic plans to hemiplegic patients. The radial extra-corporeal shock-wave therapy has promising results in patients with musculoskeletal problems and in those with various causes of HSP, including spasticity, rotator cuff problems, adhesive capsulitis, and complex regional pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age ranges from 40 to 60 years.
2. Spasticity of upper limb ranges from mild to moderate (grade 1+: 2) according to modified aschworth scale (MAS).
3. Patients with sufficient cognitive abilities that enables them to understand and follow instructions (Mini-Mental Scale >24).
4. Patient who understand the study process and signed the informed consent form.
5. Patient with stroke more than 3 months ago.

8. Patient with shoulder pain and limited range of motion (ROM) or loss of motion in the proximal arm on the hemiplegic side.

Exclusion Criteria:

* 1. Patients who cannot express their own pain intensity. 2. Patients with a history of trauma or surgery to the shoulder on the affected side.

  3. Patients with history of oral NSAIDs 3 days before this study or take warfarin medication with an international normalized ratio above 4.0.

  4. Patients with a history of shoulder pain before the stroke. 6. Patients who have received a previous shoulder intra-articular injection or other interventions on the affected shoulder within one month before rESWT.

  7. Patients with cardiac pacemaker. 8. Patients who have osteoporosis. 9. Patients with psychological problems.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
The pain pressure threshold (PPT) assessment by using pressure algometer procedures | Baseline
  Pain pressure threshold measurement will be obtained in the same order for all patients.The pressure will be applied with 0.785 cm2 rubber tip at a rate of 1 kg/cm2/sec 27 at the site of measurement. The measurement will at the mid-belly of the deltoid of the painful shoulder. The tip of the algometer will be positioned on this specific point. By pushing the algometer, the force will be applied to the mid belly of deltoid gradually increased. The patients will not allowed to see the algometer display in any moment, and, as soon as the volunteers experience a painful sensation, they say "stop", the algometer will immediately release and the force (in Kpa) will be read from the display. Pain pressure threshold will be measured three times per patient on each site and the average will be calculated and will be used for analysis.

SECONDARY OUTCOMES:
Shoulder range of motion assessment by using magnetic inclinometer | Baseline
  Total shoulder flexion will be measured with full elbow extension and leading with the thumb to ensure consistent rotation. The inclinometer will placed along the shaft of the humerus perpendicular to the plane of motion. Total shoulder abduction will be measured with full elbow extension and leading with the thumb to ensure consistent rotation. The inclinometer will placed along the shaft of the humerus perpendicular to the plane of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim A Abu-Ella, MSC, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wilson RD, Chae J. Hemiplegic Shoulder Pain. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):641-55. doi: 10.1016/j.pmr.2015.06.007. Epub 2015 Sep 9. PMID 26522903